CLINICAL TRIAL: NCT03966690
Title: Maximum Strength and Ratio of Leg Extension and Leg Flexion in Elite Soccer Players. A Comparison of an Open Versus Closed Isokinetic System
Brief Title: Rate of Leg Curl to Leg Press During Isokinetic Testing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: IMP_Test
Record Dates: First submitted 2019-05-23; First posted 2019-05-29 (Actual); Last update posted 2019-05-31 (Actual); Status verified 2019-05

CONDITIONS: Muscle Strain
MeSH Terms: conditions — Sprains and Strains

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- leg curl device starters (Experimental): Group A randomly assigned to start with legcurl device
  Interventions: Device: Isokinetic leg extension/-flexion on a legpress device; Device: Isokinetic leg extension/-flexion on a legcurl device
- legpress device starters (Experimental): Group A randomly assigned to start with legpress device
  Interventions: Device: Isokinetic leg extension/-flexion on a legpress device; Device: Isokinetic leg extension/-flexion on a legcurl device

INTERVENTIONS:
Device: Isokinetic leg extension/-flexion on a legpress device — Maximum strength and rate of leg-flexion /-extension during legpress exercise
Device: Isokinetic leg extension/-flexion on a legcurl device — Maximum strength and rate of leg-flexion /-extension during legcurl exercise

SUMMARY:
The functional condition of the leg muscles is not only relevant to performance in sports, but is also of great importance in health, prevention and rehabilitation, where not only the general strength level is decisive but also the relationship between individual muscle groups. Among other things the H-Q-ratio (strength ratio of "hamstring" muscles to quadriceps muscles) is often used to diagnose possible imbalances. Isokinetic force measurements have established themselves as the gold standard in competitive football. In this context, however, force tests in the open kinetic chain (OKC) have almost exclusively been used so far. Especially force measurements in the closed kinetic chain (CKC) could have a higher relevance regarding functionality. The H-Q-ratio should better be called the flex-ext-ratio in the CKC due to the involvement of the hip muscles. There is little data in the literature on leg force or flex-ext-ratio in CKC. In particular, there is hardly any comparative data for isokinetic measurement systems in the CKC. Using a cross over design and randomly allocating 28 competitive football players into two groups (n=14 each) that either started tests with the leg press or legcurl device, the investigators assumed (1) a significantly lower flex-ext-ratio in the CKC compared to the OKC, (2) a correlation between the isokinetic measurement systems in the OKC and the CKC, and (3) a significant superiority of the leg press to predict functional performance of the lower limbs.

ELIGIBILITY:
Inclusion Criteria:

* male elite soccer players (5th-6th German soccer division)

Exclusion Criteria:

* no acute injuries

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Male elite soccer player
Enrollment: 28 (Actual)
Dates: Start 2018-08-15 (Actual); Primary Completion 2019-02-15 (Actual); Study Completion 2019-05-15 (Actual)

PRIMARY OUTCOMES:
Leg extension/leg-flexion rate | at baseline
  Rate of leg extension to leg-flexion

SECONDARY OUTCOMES:
Isokinetic leg extensors strength | at baseline
  Maximum isokinetic strength of the leg extensors as determined by an isokinetic legpress device (Physiomed, Laipersdorf, Germany)
Isokinetic leg flexors strength | at baseline
  Maximum isokinetic strength of the leg flexors as determined by an isokinetic legpress device (Physiomed, Laipersdorf, Germany)
Y-Balance Test | at baseline
  Dynamic motor-control as determined by the Y-Balance test
Maximum jumping height | at baseline
  Maximum jumping height as determined by the counter movement jump

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Kemmler, PhD, Study Chair — Institute of Medical Physics, University of Erlangen-Nürnberg, Germany
Locations (1):
- Institute of Medical Physics, University of Erlangen-Nurnberg, Erlangen, Germany

IPD SHARING:
Plan to Share IPD: No